CLINICAL TRIAL: NCT04764409
Title: Prevention and Treatment of Complications of Endovascular Methods in Patients With Malignant Liver Tumors
Acronym: PATOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Clinical Hospital RZD-Medicine, Russian Federation (Other)
Responsible Party: Principal Investigator, Stukalova Oksana Yuryevna, Principal Investigator, Central Clinical Hospital RZD-Medicine, Russian Federation
Other Study IDs: CCHRZD00001
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hepatic Cancer; Metastatic Cancer; Chemotherapy Effect
Keywords: Chemoembolization
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: This group includes patients who underwent chemoembolization of hepatic arteria
  Interventions: Procedure: Chemoembolization
- Group 2: This group includes patients who underwent chemoinfusion of hepatic arteria
  Interventions: Procedure: Chemoinfusion

INTERVENTIONS:
Procedure: Chemoembolization — Transarterial Chemoembolization (TACE)
  Groups: Group 1
Procedure: Chemoinfusion — Transarterial Infusion (TAI)
  Groups: Group 2

SUMMARY:
In the structure of malignant liver lesions, two main groups are distinguished - primary liver cancer and metastatic liver damage. The five-year survival rate of patients with malignant liver tumors does not exceed 6%. The main and radical method of treatment today is liver resection. However, surgical treatment is possible only in 10-25% of patients. At the same time, recurrence of malignant tumors is observed in 60-80% of cases within five years after surgery, and the number of candidates for repeated liver resection does not exceed 10%. The high toxicity of systemic chemotherapy limits its use in this group of patients. In this connection, minimally invasive and at the same time effective methods of local treatment of malignant liver tumors have been introduced into clinical practice. These methods include: hepatic artery chemoinfusion, chemoembolization and oil chemoembolization.

Currently, a large world experience has already been accumulated in the application of the above methods of treatment. However, any, even minimally invasive, surgical manipulation can be associated with the development of complications of varying severity. If complications arise, there is a risk of interruption of palliative care, which entails a significant reduction in life expectancy. According to domestic and foreign literature, the occurrence of complications after intra-arterial chemoembolization occurs in 0.4-10% of patients, and after intra-arterial chemoinfusion - in 5-30% of patients. In the overwhelming majority of scientific works, the description of the complications that have arisen is reduced to listing the latter. Currently, in the Russian and foreign scientific literature there is no systematization of complications, there is no single clinical classification, algorithms for the prevention and treatment of complications arising after local intravascular methods of treatment of patients with malignant liver tumors.

The study and systematization of complications arising after intra-arterial chemoembolization and chemoinfusion of the hepatic artery in patients with malignant liver tumors will make it possible to create prevention and treatment algorithms. Thus, it will help prevent interruption of palliative care and increase the life expectancy of this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years old;
2. Histologically confirmed diagnosis of liver cancer or metastatic liver disease;
3. Patients who have not received systemic antitumor therapy within the last 6 months

Exclusion Criteria:

1. Metachronous (within 3 years) or synchronous other oncological disease with the exception of healed carcinoma in situ;
2. The volume of liver damage according to computed tomography is more than 60%;
3. Increase in the level of transaminases by more than 2 times;
4. The level of bilirubin is more than 50 μmol / l;
5. Heart failure stage II B-III, Functional Class III-IV;
6. The presence of uncorrected coagulopathy;
7. Renal failure stage III-IV;
8. Ascites 2-3 degrees;
9. The general condition of the patient is below 60% on the Karnofsky index and above 2 points on the Eastern Cooperative Oncology Group (ECOG) scale;
10. Liver damage - more than 7 points on the Child-Pugh scale;
11. Damage to the central nervous system;
12. Anemia of severe severity;
13. Pregnancy;
14. Active autoimmune disease;
15. Presence of HIV infection, active forms of tuberculosis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned to include patients with primary liver cancer and metastatic liver disease, after chemoembolization or chemoinfusion of the hepatic artery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Identification of all the kinds of complications according to the Common Terminology Criteria for Adverse Events (CTCAE v4.0) and their systematization. | 2 years
  This systematization will lead to the creation of algorithms of prevention and treatment of complications of endovascular methods in patients with malignant liver tumors. For the assessment of the severity of complications there will be created a new scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Clinical Hospital RZD-Medicine, Russian Federation, Moscow, Moscow's Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes